CLINICAL TRIAL: NCT02703519
Title: Optimierung Der Uterotomie-Wundheilung Nach Re-Sectio Caesarea
Brief Title: Optimization of the Healing Process of the Uterine Scar Tissue After Re-cesarean Section
Acronym: OPSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Otto-von-Guericke University Magdeburg (Other)
Responsible Party: Principal Investigator, Gregor Seliger, Dr. med., chief resident, Martin-Luther-Universität Halle-Wittenberg
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OPSTAR
Record Dates: First submitted 2016-03-06; First posted 2016-03-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Scar; Previous Cesarean Section; Complications; Cesarean Section, Wound, Dehiscence
Keywords: cesarean section, repeat; uterine scar tissue; transvaginal ultrasound; uterine rupture; placenta accreta; placenta percreta; placenta increta
MeSH Terms: conditions — Cicatrix; Wounds and Injuries; Uterine Rupture; Placenta Accreta

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 cesarean section (No Intervention): control group
- 2 cesarean sections (No Intervention): control group
- resection of uterine scar tissue (Experimental): 2 cesarean sections with resection of uterine scar tissue from first cesarean section
  Interventions: Procedure: resection of uterine scar tissue

INTERVENTIONS:
Procedure: resection of uterine scar tissue — resection of uterine scar tissue of a previous cesarean section during a second cesarean section
  Arms: resection of uterine scar tissue

SUMMARY:
This prospective, controlled, clinical, intervention study measures the number of uterine Cesarean section scars and median myometrial thickness of women who underwent two Cesarean sections six to nine months after their last Cesarean section using transvaginal ultrasound.

It is the purpose of the study to assess if a resection of the uterine scar from a previous Cesarean section during a second Cesarean section could lead to a decrease in risk for subsequent pregnancies.

DETAILED DESCRIPTION:
The average number of Cesarean sections in Germany has doubled from 1991 to 2011, making up 32,1% of all deliveries in 2011.

Several studies describe instances in which pregnancies following a previous Cesarean section were accompanied by complications such as life-threatening bleeding, placenta previa, placenta accreta, increta or percreta and dehiscence or uterine rupture.

The risk of those complications increases further with the uterine scar tissue of a second Cesarean section.

Today it is already common practice to resect uterine scars if the scar of a previous Cesarean section becomes symptomatic, or when a non-symptomatic uterine rupture or serious dehiscence are discovered during a Cesarean delivery.

In this study all participants of the interventional group are examined via intraoperative ultrasound to identify the first uterine Cesarean section scar and resect it completely.

Six to nine months after the resection participants will return for a one time follow-up. At this time, the investigators will measure the number of uterine scars and median myometrial thickness using transvaginal ultrasound. The results will be compared with those of two control groups, consisting of women who underwent either one or two Cesarean sections without the intervention.

The aim of the present study is to asses if the number of uterine scars and median myometrial thickness can be improved by the resection of the first uterine scar during a subsequent Cesarean section.

This will allow the investigators to draw conclusions regarding the benefit of routine resections of uterine Cesarean section scars, and whether this practice could lead to a decreased risk for women undergoing two or more Cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* primary or secondary indication for cesarean section 6 to 9 months prior to the examination date

Exclusion Criteria:

* <18 years old
* current pregnancy
* congenital deformity of the uterus
* former surgery of the uterine myometrium

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
number of uterine Cesarean section scars using transvaginal ultrasound | 6-9 months

SECONDARY OUTCOMES:
median myometrial thickness of lower uterine segment using transvaginal ultrasound | 6-9months

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Seliger, Dr. med., Principal Investigator — Maternity Clinic/Perinatal Treatment Center, Halle University Hospital, Martin-Luther-Universität Halle-Wittenberg; Michael Tchirikov, Prof., Study Chair — Maternity Clinic/Perinatal Treatment Center, Halle University Hospital, Martin-Luther-Universität Halle-Wittenberg; Serben-Dan Costa, Prof., Principal Investigator — Maternity Clinic, Magdeburg University Hospital
Locations (2):
- Germany (2):
  - Maternity Clinic/Perinatal Treatment Center, Halle University Hospital, Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
  - Maternity Clinic, Magdeburg University Hospital, Magdeburg, Saxony-Anhalt

IPD SHARING:
Plan to Share IPD: No